CLINICAL TRIAL: NCT05446610
Title: Development of a Novel Functional Food Enriched With Beta-glucans Isolated From Edible Mushrooms of Greek Habitats
Brief Title: Investigating Effects in Intestinal Permeability of Rich in Beta-glucans Pleurotus Eryngii Mushrooms Fermentation Supernatants: an Ex-vivo Study
Acronym: FUNglucan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Harokopio University (Other); Agricultural University of Athens (Other); National Hellenic Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T1EDK-03404
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: paracellular permeability; transcellular permability; Pleurotus eryngii; beta glucan; prebiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gut barrier function treatments (Experimental): Stressor, fibre, combination of treatments.
  Interventions: Other: Fermented product of Pleurotus eryngii mushroom

INTERVENTIONS:
Other: Fermented product of Pleurotus eryngii mushroom — I Stimulation of human colonic biopsies with the fermented product of Pleurotus eryngii mushroom

SUMMARY:
The aim of the present study was to investigate the ability of Pleurotus eryngii mushrooms fermentation products (FS) to counteract induced intestinal hyperpermeability in human colonic tissues in an ex vivo system.

DETAILED DESCRIPTION:
Collection of colon biopsies through sigmoidoscopy procedure will take place and the collected biopsies will be mounted in Ussing Chambers. Already collected fermentation supernatants will be added to the mucosal side of the biopsy together with a stressor and two permeability markers, in order to investigate the effects of the fibre fractions on both paracellular and transcellular permeability.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent prior to any study related procedures
2. Age 18-65 years
3. Willing to abstain from regular consumption of prebiotics/probiotics products or medication known to alter gastrointestinal functions at least 4 weeks prior to the study visits

Exclusion Criteria:

1. Previous complicated gastrointestinal surgery
2. Presence of gastrointestinal disorder or any disorder which the principal investigator considers to affect the results of the study
3. Current diagnosis of psychiatric disease
4. Current and past diagnosis inflammatory gastrointestinal disease (e.g. Irritable Bowel Disease)
5. Systemic use of antibiotics or steroids medications in the last 3 months
6. Frequent use of NSAID (Non Steroidal Anti Inflammatory Drugs) the last 2 months prior to study visits
7. Regular consumption of prebiotic/probiotic products for the past 4 weeks
8. Abuse of alcohol or drugs
9. Frequent use of laxatives, anti-diarrheal, anti-cholinergic within last 12 weeks prior to study visits
10. Pregnancy and breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline of barrier function (paracellular permeability) after 90 minutes of ex vivo stimulation of the colonic biopsies. | Barrier function will be measured at baseline and after 90 minutes of ex vivo stimulation of the colonic biopsies.
  Barrier function (paracellular permeability) will be evaluated with the use of marker related this permeability, through immunofluoresence.
Change from baseline of barrier function (transcellular permeability) after 90 minutes of ex vivo stimulation of the colonic biopsies. | Barrier function will be measured at baseline and after 90 minutes of ex vivo stimulation of the colonic biopsies.
  Barrier function (transcellular permeability) will be evaluated with the use of marker related to this permeability, through ELISA tecnhique.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Rangel, As.Professor, Principal Investigator — Örebro University, School of Medical Sciences, Sweden
Locations (1):
- Campus USÖ, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitsou EK, Saxami G, Stamoulou E, Kerezoudi E, Terzi E, Koutrotsios G, Bekiaris G, Zervakis GI, Mountzouris KC, Pletsa V, Kyriacou A. Effects of Rich in Beta-Glucans Edible Mushrooms on Aging Gut Microbiota Characteristics: An In Vitro Study. Molecules. 2020 Jun 18;25(12):2806. doi: 10.3390/molecules25122806. PMID 32570735
- [Result] Boulaka A, Christodoulou P, Vlassopoulou M, Koutrotsios G, Bekiaris G, Zervakis GI, Mitsou EK, Saxami G, Kyriacou A, Zervou M, Georgiadis P, Pletsa V. Genoprotective Properties and Metabolites of beta-Glucan-Rich Edible Mushrooms Following Their In Vitro Fermentation by Human Faecal Microbiota. Molecules. 2020 Aug 4;25(15):3554. doi: 10.3390/molecules25153554. PMID 32759726
- [Result] Saxami G, Kerezoudi EN, Mitsou EK, Koutrotsios G, Zervakis GI, Pletsa V, Kyriacou A. Fermentation Supernatants of Pleurotus eryngii Mushroom Ameliorate Intestinal Epithelial Barrier Dysfunction in Lipopolysaccharide-Induced Caco-2 Cells via Upregulation of Tight Junctions. Microorganisms. 2021 Oct 1;9(10):2071. doi: 10.3390/microorganisms9102071. PMID 34683391
- See also: Research center website — https://www.oru.se/english/research/research-environments/mh/nutrition-gut-brain-interactions-research-centre-ngbi/
- See also: Description Project's official website — https://funglucan.hua.gr/
- See also: Description Project's official facebook website — https://www.facebook.com/FUNglucan-2604410072963486/
- See also: Description Project's official instagram website — https://www.instagram.com/funglucan/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT05446610/Prot_SAP_000.pdf